CLINICAL TRIAL: NCT04737681
Title: Influence of Body Weight and Composition on Immune Recovery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 19-26HC
Record Dates: First submitted 2020-08-24; First posted 2021-02-04 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: BMI/Body Composition
MeSH Terms: interventions — Body Composition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal BMI: BMI 18.5-24.9 kg/m2
  Interventions: Other: body composition
- Obese BMI: BMI ≥ 30 kg/m2
  Interventions: Other: body composition

INTERVENTIONS:
Other: body composition — This is an observational study to determine immune response and skin barrier restoration in individuals with and without obesity.

SUMMARY:
Immune dysfunction in individuals with obesity, secondary to chronic inflammation, may have an acute impact on War fighter health and readiness, and subsequent lethality. Indeed, ~51% of military personnel ages 17 or older are overweight, and ~15% have obesity (ranging from 6.4% in the Marine Corps to 18.0% in the Army). In conjunction with in vitro functional tests to assess systemic immune function, the suction blister model is a minimally invasive procedure that allows in vivo assessment of immune function (i.e., skin barrier restoration), and related mechanisms (i.e., pro- and anti-inflammatory cytokine responses at the wound site during the early phases of wound healing), consequent to obesity. We have demonstrated that the blister wound model reliably assesses skin barrier restoration and immune function at the wound site; and that relatively modest sleep disruption degrades immune response at the site of the disrupted skin barrier and delays the initial restoration of the skin barrier. However, our prior work excluded participants with obesity (≥30 kg/m2), since obesity is associated with an altered inflammatory response which may subsequently impact the body's functional response to a skin wound. Prior studies have indicated that immune function and wound healing is perturbed in individuals with obesity versus those without obesity. Existing research mainly relied on blood biomarkers and in vitro tests to assess systemic immune function; however, incorporating the blister wound model permits evaluation of the functional immune response to obesity in addition to local immune response at the wound site. Further, military personnel with obesity may be more physically active than civilians with obesity, which could mitigate the effects of obesity on immune dysfunction. Therefore, the primary aim of this parallel-group study is to utilize a suction blister model and in vitro functional assays to examine differences in immune function between participants without obesity (BMI 18.5-24.9 kg/m2) and with obesity (BMI ≥ 30 kg/m2) and related mechanisms (e.g., local cytokine response at the wound site and circulating markers of inflammation). Research will be conducted in a laboratory environment using males and females with obesity (BMI ≥ 30 kg/m2) compared to normal weight (BMI 18.5-24.9 kg/m2) controls. Participants in the study described herein (n = 50; n = 25 with obesity and n = 25 lean) will undergo baseline testing and a period of dietary surveillance prior to induction of up to eight blisters via suction on participant's forearm, after which time the top layer of blisters will be removed to reveal the dermal layer of skin. The primary outcome measure is initial restoration of the skin barrier (via transepidermal water loss) and additional outcome measures include immune function (e.g., circulating markers of inflammation, cytokines at the blister site, and secretory immunoglobin) and nutrient status. Additionally, to assess the impact of BMI on skeletal muscle inflammation, a subset of volunteers (n = 12 with obesity and n =12 lean) will undergo a single muscle biopsy at the conclusion of skin barrier restoration. Findings from this study will determine if obesity affects the early phases of wound healing and whether further study is warranted, e.g., do stressors exacerbate immune decrements observed in obese individuals, or can nutrition counter-measures mitigate immune decrements given that micronutrient deficiency is common in individuals with obesity.

DETAILED DESCRIPTION:
See brief summary above.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18 (or 17 for military personnel) and 39 (i.e., consistent with the age range of 95% of Active Duty enlisted and 75% of Active Duty officers)
* Have a Body Mass Index (BMI) in the range of 18.5 to <25 kg/m2 and have a percent body fat by circumference measurements that meets the Army's max allowable body fat standards for individuals classified as "without obesity"; or have a BMI ≥ 30 kg/m2 and have a percent body fat by circumference measurements that exceeds the Army's max allowable body fat standards for individuals classified as "with obesity" (40).
* Have been weight stable (+/- 5 lbs.) for the past two months (not including temporary body weight fluctuations due to menstrual cycle) and agree not to attempt to lose or gain weight for the duration of the study;
* Participate in 120-300 mins of aerobic exercise over the course of at least 3 days per week as indicated by self-report data and confirmed during the study via actigraphy (i.e., consistent with the self-reported exercise habits of a majority of active duty military personnel) (1, 41)
* Are willing to participate in all study procedures and comply with all study instruction.
* Females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or able to provide documentation of oral/hormonal contraceptive use which contains low-dose estrogen/progesterone to maintain continuous levels throughout the 28-day cycle (i.e., no placebos)
* Pass a general medical clearance.

Exclusion Criteria:

* have a tattoo on both forearms that obscures the forearms and doesn't allow space for the suction blister induction;
* experienced more than a ~5 lbs. weight gain or loss in the last month than is not transient (e.g., menstrual).
* participate in more than 300 minutes of aerobic exercise per week as indicated by self-report data and confirmed during the study via actigraphy (i.e., consistent with self-reported exercise habits of ~20% of active duty military personnel) (1, 41).
* are habitually taking nonsteroidal anti-inflammatory drugs (e.g., Advil), aspirin, lipid-lowering drugs, corticosteroids or immunosuppressants (e.g. Humira);
* are immune-compromised (e.g., chemotherapy or radiation treatment);
* are suffering from an autoimmune disease (e.g., lupus);
* recovering from a surgery within the past 6 months;
* Current doctor-diagnosed and/or treated diabetes, hypertension or dyslipidemia
* are suffering from sleep apnea;
* smoke, dip, chew or vape tobacco or nicotine-containing products.
* regularly (more than 2 days per week) sleep less than 7 hours or more than 9 hours per night; or, take a nap 3 or more days per week.
* Pregnant or lactating
* problems with blood clotting (in the subset of participants receiving muscle biopsies only)
* allergy to lidocaine (in the subset of participants receiving biopsies only)

Females Only:

• Have abnormal menstrual cycles (not between 26-32 days in duration; or not 5-6 menstrual cycles within the past 6 month) or those that have had an intrauterine device (IUD) placed with the last month or removed within the past 3 months.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participant population will consist of military personnel (male or female) and civilians. Participants will be matched for both sex and the proportion of participants above and below 30 years of age. Potential participants will be screened for body mass index (BMI), percent body fat and aerobic exercise habits.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Initial restoration of the skin barrier | 4-10 days
  initial restoration of the skin barrier (via transepidermal water loss)

SECONDARY OUTCOMES:
circulation markers of inflammation | baseline
  Interleukin (IL) 6, IL8, tumor necrosis factor alpha, c-reactive protein
cytokines at the wound site | 72 hours
  Interleukin (IL) 6, IL8, IL10, tumor necrosis factor alpha
mucosal immune function | baseline
  mucosal immune function will be measured via salivary secretory immunoglobulin A

OTHER OUTCOMES:
nutrient status | baseline
  vitamin C, iron and vitamin D status measured from blood

CONTACTS AND LOCATIONS:
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No